CLINICAL TRIAL: NCT02683538
Title: Radiofrequency Ablation Using Octopus Electrodes for Treatment of Focal Liver Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0364
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma; Metastasis; Cholangiocarcinoma
Keywords: RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Separable cluster electrode (Experimental): radiofrequency ablation (RFA) using separable cluster electrode in switching monopolar mode.
  Interventions: Device: Separable cluster electrode (Octopus®)

INTERVENTIONS:
Device: Separable cluster electrode (Octopus®) — Patients undergo RFA under ultrasound guidance, and separable cluster electrodes are used for RFA in monopolar switching mode, using multiple overlapping technique to create larger ablative zones.

SUMMARY:
The purpose of this study is to evaluate the clinical feasibility and short-term outcome of switching monopolar RFA using a separable cluster electrode in patients with primary and secondary liver malignancies.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is one of minimal invasive treatment methods and it has been showing comparable overall survival with surgery in early or small hepatocellular carcinomas (HCCs) and better cost-effectiveness. However, it is suffering from high local tumor progression (LTP) rate. To reduce LTP rate, creation of large ablative zone has been attempted in various strategies. A separable cluster electrode is a new type of RFA electrode. It consists of three individual applicators and the applicators can be incorporated as a single handle such as a cluster electrode, and can be separated as three electrodes, depending on operators' needs. It allows high flexibility to operators and the preclinical results were promising. Herein, we want to evaluate the clinical feasibility of the electrodes by observing major complication rates, technical success rate and 12-months LTP rate.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic malignancies diagnosed on biopsy OR
* Typical imaging features of hepatocellular carcinoma (HCC) on computed tomography (CT) or magnetic resonance imaging (MRI) according to AASLD guideline
* Typical imaging feature of metastasis on CT or MRI AND
* 1~5 tumors equal to or smaller than 5cm in the liver
* no direct contact with or invasion into the hepatic hilar structures or inferior vena cava (IVC)
* Eastern Cooperative Oncology Group performance status of 0
* Patients who signed informed consent

Exclusion Criteria: Patients with any of followings are excluded.

* Patients with uncontrolled coagulopathy
* Patients with Child-Pugh classification C
* Patients with tumor invasion in major portal vein or hepatic vein branch
* Extrahepatic metastasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Major complication rate after Radiofrequency ablation (RFA) | 30 days after RFA
  Rates of major complication according to Society of Interventional Radiology (SIR) grading system, which refers to an event that leads to substantial morbidity and disability (SIR classification C-E).

SECONDARY OUTCOMES:
Technical success | 1 day after RFA
  Technical success addresses that the tumor was treated according to protocol and completely covered by ablative zone on pre-RFA image and post-RFA image side-by-side comparison.
Local control rate | 12 months after RFA
  Rate of local tumor progression after RFA

OTHER OUTCOMES:
total procedure time | 1 day after RFA
  total procedure time per patients was recorded.
Ablative zone volume | 1 day after RFA
  ablative zone volume measurement for each tumor on post-RFA cross sectional imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No